CLINICAL TRIAL: NCT03906760
Title: Bladder Endometriosis: Evaluation in MRI of the Involvement of the Posterior Inferior Wall
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 17-171
Record Dates: First submitted 2018-11-15; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Endometrial Bladder Disease
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Magnetic resonance imaging (MRI) — MRI protocol associating sagittal and axial (+/- coronal) sequences in T2 + / - turbo spin T1 weighting with fat saturation.

SUMMARY:
Evaluate MRI criteria for involvement of the posterior inferior wall of the bladder in patients with endometrial bladder disease.

DETAILED DESCRIPTION:
PURPOSE: to retrospectively evaluate on MRI the local staging with assessment of ureteral orifices extension in bladder endometriosis./ MATERIALS AND METHODS: Institutional review board approval for this study was obtained and waived written informed consent. The MR images of 39 patients operated for bladder endometriosis over a 6 years period in 3 university Lyon hospitals were reviewed. Two experienced readers reported the vesical repletion volume, the largest lesion size, the location and extension of the lesion within the bladder wall, the distance between the ureteral orifices and the lesion when the vesicovaginal wall was involved, the presence of muco-sub mucosal complex edema and the association with external adenomyosis. MR images were compared with surgical and pathological findings. Efficacy parameters were calculated with 95% confidence interval (CI).

ELIGIBILITY:
Inclusion Criteria:

* Patient operated for pelvic endometriosis with bladder resection.
* Performing a preoperative pelvic MRI with at least 2 perpendicular T2 planes

Exclusion Criteria:

* Refusal to use clinical data and exploration acquired
* Absence of interpretable preoperative pelvic MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients treated in the gynecological surgery departments of the University Hospital Center of the Civil Hospitals of Lyon: Lyon Sud.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of MRI data with intraoperative data and anatomopathology. | Through bladder endometriosis surgery
  A bladder lesion will be retained when a signal abnormality is present on at least two different sectional planes or weights. The topography of the lesion will be related to the vesico-uterine cul-de-sac, its lateralization, its distance from the bladder neck and meatus, its size and its signal.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud -Service de Radiologie, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No